CLINICAL TRIAL: NCT01797016
Title: Comparing Blood Count Test Measures to Flow Cytometry in Healthy Patients to Acute General Syndrome Patients
Brief Title: Platelet Leukocyte Aggregates in Acute Cardiac Syndrome vs Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Najib Dally, Head of Hematology Institute, Ziv Hospital
Other Study IDs: 0059-12-ZIV
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; flow cytometry; Blood Cell Count; Platelet Activation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project aims to refine previous studies including the investigators work recently published in August 2012 Journal Thrombosis and Thrombolysis. That study showed a relationship between the level of platelet leukocyte aggregates in patients with acute coronary syndrome. The investigators intend to compare the characteristics of platelets, monocytes and neutrophil data of volume, scatter and conductivity obtained from routine blood count level with flow cytometry results defining platelet leukocyte aggregates. The investigators hypothesize that there will be a direct correlation between elevated platelet-leukocyte aggregates and biophysical data from the blood count.

DETAILED DESCRIPTION:
The goal is to investigate whether there is a simple and inexpensive method to test the level of platelet leukocyte aggregates through the blood count test. The parameters which are obtained routinely for white blood cell counts include: capacity - electrical conductivity (conductivity) - dispersion (scatter), and volume. Though these values are not reported routinely, they can be accessed for each blood count.

The premise is that through blood counts (no need for specialized flow cytometry) and through the parameters mentioned a conclusion can be reached about platelet leukocyte aggregates. This will then aid in prognosis about the risk of an acute event for every patient with ischemic heart disease who comes to the emergency room.

ELIGIBILITY:
Inclusion Criteria:Signed consent form, over 18 years of age, diagnosis of STEMI or non-STEMI as per following:

* Acute ST Elevation Myocardial Infarction (STEMI) was diagnosed in patients with high level of troponin I (>0.4 ng/ml), ST segment elevation in at least two contiguous leads of the ECG (or new LBBB) and/or ischemic chest pain.
* Acute Non ST Elevation Myocardial Infarction (Non STEMI) was diagnosed if level of troponin I was > 0.4 ng/ml, patient had ischemic chest pain or ST-T depression and/or T-wave inversion on ECG.

Exclusion Criteria:Inability to sign consent form, under 18, participation in other research projects within previous 6 months.

-

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute Myocardial Infact
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Detection of platelet-leukocyte aggregates by routine blood count. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nagib Dally, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel